CLINICAL TRIAL: NCT03108014
Title: Beginnings Study Follow up
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206291
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast milk fed: Fed primarily breast fed as an infant
- Cow's Milk based infant formula fed: Fed primarily cow's milk based infant formula for the first year of life
- Soy-protein based formula fed: Fed primarily soy-protein based infant formula during the first year of life

SUMMARY:
This study will help us learn more about how early infant diet may influence child's growth and development at age 14.

DETAILED DESCRIPTION:
This study is to follow the infants that were enrolled in Beginnings study which purpose was to characterize physical growth, body composition, dietary intake, neurobehavioral development, and brain function of infants and children fed mostly breast milk, milk based formula, or soy based formula during their first year of life up to age 6. This study will call back those children when they turn 14 to compare growth, sexual maturation, and development between the three diets.

ELIGIBILITY:
Inclusion Criteria:

* Beginnings study former participants

Exclusion Criteria:

* Dropped participants for medical diagnosis or medical conditions

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Former Beginnings participants between ages 13 and 15 years
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Growth and development | 14 years
  Will be determined with body composition equipment

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, RD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No